CLINICAL TRIAL: NCT03009110
Title: Prophylactic Negative Pressure Wound Therapy in Obese Women at Cesarean: a Multicenter Randomized Trial
Brief Title: Preventing Adverse Incisional Outcomes at Cesarean Multicenter Trial
Acronym: Prevena-C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation following interim analysis
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); 3M (Industry)
Responsible Party: Principal Investigator, David Haas, Professor of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB ID #: 201603062; 1R01HD086007-01A1 (NIH)
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Surgical Wound Infection; Cesarean Section
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prophylactic NPWT (Experimental): Women assigned to prophylactic NPWT will have the Prevena device applied and secured with fixation adhesion strips. The device will be monitored while the patient is in the hospital to confirm that it is functioning well. The device will be removed prior to discharge, typically on postoperative day 4, but longer for up to 7 days for patients who remain hospitalized.
  Interventions: Device: Prophylactic NPWT
- Standard Dressing (Active Comparator): Women assigned to standard care will receive routine postoperative wound dressing consisting of layers of gauze and adhesive tap. The dressing will be removed after 24 - 48 hours.
  Interventions: Device: Standard Dressing

INTERVENTIONS:
Device: Prophylactic NPWT — The Prevena NPWT system is a small, lightweight, portable suction device consisting of an electric motor-driven vacuum pump connected to a proprietary foam and adhesive dressing. It is supplied as a pump with a sterile dressing kit and two batteries. Different dressing sizes are available for transverse and vertical incisions ranging from 13 to 20 cm and more. The pump maintains negative pressure of -125 mmHg to the wound surface. The device is placed after skin closure.
  Other Names: Prevena
  Arms: Prophylactic NPWT
Device: Standard Dressing — Standard wound dressing is routine postoperative wound dressing consisting of layers of gauze and adhesive tape.
  Arms: Standard Dressing

SUMMARY:
The Prophylactic Negative Pressure Wound Therapy in Obese Women at Cesarean Trial is a large pragmatic multi-center randomized clinical trial designed to evaluate the effectiveness, safety and cost-effectiveness of prophylactic negative pressure wound therapy (NPWT) - a closed, sealed system that applies negative pressure to the wound surface via a single-use, battery-powered, portable device - to decrease surgical site infections (SSIs) in obese women.

DETAILED DESCRIPTION:
Experimental evidence suggests that NPWT promotes wound healing by removing exudate, approximating the wound edges, and reducing bacterial contamination. Obesity (body mass index [BMI] ≥30kg/m2) increases the risk for both cesarean delivery and SSIs compared to non-obese women. The increased risk of SSIs is in part due to the increased thickness of the subcutaneous space, allowing collection of exudates and increasing tension on wound edges, promoting the growth of bacteria, and leading to wound infection and breakdown. Thus, prophylactic NPWT may be particularly effective in this patient population.

During the 5-year project period, investigators from 4 collaborating perinatal centers in the United Stated (two university and two community) will randomize 2850 obese women undergoing cesarean delivery to receive either prophylactic negative pressure wound therapy with the Prevena device or standard wound dressing. Women will be followed up to 30 days postoperatively to ascertain study outcomes.

The primary outcome for the trial is superficial or deep SSI after cesarean according to the CDC's National Healthcare Safety Network definitions. The investigators will also assess other wound complications, adverse events potentially attributable to NPWT and cost-effectiveness as measured by incremental cost per case of SSI prevented and per quality-adjusted life year (QALY).

ELIGIBILITY:
Inclusion Criteria

* Gestational age ≥23weeks
* BMI≥30 Pre-pregnancy or BMI at first prenatal visit
* Planned or unplanned cesarean delivery

Exclusion Criteria:

* Non-availability for postoperative follow-up
* Contraindication to NPWT applicable to women undergoing cesarean: Pre-existing infection around incision site, Bleeding disorder, Therapeutic anticoagulation, Irradiated skin, Allergy to any component of the dressing (e.g. silver, acrylic, silicone, adhesive tape)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1624 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Methodius G Tuuli, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (6):
- United States (6):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Eskenazi Hopsital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Mercy Hosptial St Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mark KS, Alger L, Terplan M. Incisional negative pressure therapy to prevent wound complications following cesarean section in morbidly obese women: a pilot study. Surg Innov. 2014 Aug;21(4):345-9. doi: 10.1177/1553350613503736. Epub 2013 Sep 20. PMID 24056202
- [Background] Swift SH, Zimmerman MB, Hardy-Fairbanks AJ. Effect of Single-Use Negative Pressure Wound Therapy on Postcesarean Infections and Wound Complications for High-Risk Patients. J Reprod Med. 2015 May-Jun;60(5-6):211-8. PMID 26126306
- [Background] Bullough, L, Wilkinson, D., Burns, S, Wan, L, Changing wound care protocols to reduce postoperative caesarean section infection and readmission, Wounds , 2014 (10), 1 : 72 - 76. 46
- [Background] Chaboyer W, Anderson V, Webster J, Sneddon A, Thalib L, Gillespie BM. Negative Pressure Wound Therapy on Surgical Site Infections in Women Undergoing Elective Caesarean Sections: A Pilot RCT. Healthcare (Basel). 2014 Sep 30;2(4):417-28. doi: 10.3390/healthcare2040417. PMID 27429285
- [Derived] Tuuli MG, Liu J, Tita ATN, Longo S, Trudell A, Carter EB, Shanks A, Woolfolk C, Caughey AB, Warren DK, Odibo AO, Colditz G, Macones GA, Harper L. Effect of Prophylactic Negative Pressure Wound Therapy vs Standard Wound Dressing on Surgical-Site Infection in Obese Women After Cesarean Delivery: A Randomized Clinical Trial. JAMA. 2020 Sep 22;324(12):1180-1189. doi: 10.1001/jama.2020.13361. PMID 32960242

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prophylactic NPWT | Standard Dressing
Started | 816 | 808
Completed | 806 | 802
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic NPWT | Standard Dressing | Total
Number analyzed (Participants) | 806 | 802 | 1608
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 6
  Between 18 and 65 years | 805 | 797 | 1602
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (5.6) | 30.1 (5.9) | 29.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 806 | 802 | 1608
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 27 | 61
  Not Hispanic or Latino | 772 | 775 | 1547
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 453 | 452 | 905
  White | 331 | 330 | 661
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 20 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 806 | 802 | 1608
BMI [Mean (Standard Deviation); unit: kg / m^2] — body mass index (kg/m^2)
  kg / m^2 | 39.6 (7.7) | 39.5 (8.1) | 39.6 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Superficial or Deep Surgical Site Infections (SSIs)
Description: As defined according to the Center for Disease Control and Prevention's (CDC) National Healthcare Safety Network criteria.
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 29 | 27

2. Secondary Outcome: Number of Participants With Superficial, Deep or Organ Space SSIs (Individual Types of SSIs)
Description: As defined according to the CDC's National Healthcare Safety Network criteria.
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 29 | 27

3. Secondary Outcome: Number of Participants With Organ Space SSIs (Endometritis, Intraabdominal Abscess)
Description: As defined according to the CDC's National Healthcare Safety Network criteria.
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 2 | 2

4. Secondary Outcome: Number of Participants With Wound Hematoma, Seroma, Separation (Other Wound Complications)
Description: Frequency of wound hematoma, seroma, separation (other wound complications). Hematoma, seroma, separation (2cm or more).
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 21 | 25

5. Secondary Outcome: Number of Participants With a Composite of Any Wound Complication Including SSI, Hematoma, Seroma, Separation (2cm or More).
Description: Frequency of a composite of any wound complication including SSI, hematoma, seroma, separation (2cm or more). SSI, hematoma, seroma, separation (2cm or more).
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 52 | 54

6. Secondary Outcome: Patient Pain Score
Description: On a scale of 0 (least) - 10 (most).
Time Frame: At discharge, an average of 4 days postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
score on a scale | 3 [0 to 5] | 3 [0 to 5]

7. Secondary Outcome: Patient Pain Score
Description: On a scale of 0 (least) - 10 (most).
Time Frame: At postoperative day 30
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
score on a scale | 0 [0 to 2] | 0 [0 to 2]

8. Secondary Outcome: Patient Satisfaction Score
Description: On a scale of 0 (least) - 10 (most).
Time Frame: At discharge, an average of 4 days postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
score on a scale | 10 [8 to 10] | 9 [7 to 10]

9. Secondary Outcome: Patient Satisfaction Score
Description: On a scale of 0 (least) - 10 (most).
Time Frame: At postoperative day 30
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
score on a scale | 10 [9 to 10] | 10 [8 to 10]

10. Secondary Outcome: Number of Participants With Physician Office Visit, Emergency Room Visit, Attendance at Wound Clinic, Use Antibiotics, Hospital Readmission for Wound Related Problems (Measures of Healthcare Resource Utilization)
Description: Frequency of physician office visit, emergency room visit, attendance at wound clinic, use antibiotics, hospital readmission for wound related problems (measures of healthcare resource utilization).
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 130 | 132

11. Secondary Outcome: Number of Participants With Skin Blistering, Erythema, Wound Bleeding (Measures of Adverse Skin Events)
Description: Frequency of skin blistering, erythema, wound bleeding (measures of adverse skin events).
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prophylactic NPWT | Standard Dressing
Number analyzed (Participants) | 806 | 802
Participants | 46 | 5

12. Other Pre Specified Outcome: Types and Frequency of Different Bacteria Including Methicillin-resistant Staphylococcus Aureus
Description: Types and frequency of different bacteria including methicillin-resistant Staphylococcus aureus.
Time Frame: 30 days postoperatively
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Incremental Cost Per SSI Prevented
Description: Based on economic analysis to be done along side trial. Results of the economic analysis will be published separately from the effectiveness and safety data.
Time Frame: 30 days postoperatively
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Incremental Cost Per Quality-Adjusted Life-year
Description: as for outcome 13
Time Frame: 30 days postoperatively
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Risk Factors for Surgical Site Infections in Obese Women
Description: Based on combined cohort. Results of the risk factor analysis will be published separately from the effectiveness and safety data.
Time Frame: 30 days postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Description: Occurring within data collection period, to be reported within 24 hours of learning of the event:
  Serious Adverse Events - Death or Life-threatening situations:
  Postpartum hysterectomy for infection control Maternal sepsis Necrotizing fasciitis Maternal ICU admission
  Abnormal findings in labs or assessments will not be reported as adverse events.
  Adverse Events of special interest will be reported - mild/moderate reactions:
  Skin blisters Wound bleeding Allergic skin reaction
Arm/Group | Prophylactic NPWT | Standard Dressing
All-Cause Mortality (participants affected / at risk) | 0/806 | 0/802
Serious Adverse Events (participants affected / at risk) | 4/806 | 5/802
Other Adverse Events (participants affected / at risk) | 56/806 | 5/802
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic NPWT (N=806) | Standard Dressing (N=802)
Maternal ICU admission (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Maternal Sepsis (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Postpartum hysterectomy (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylactic NPWT (N=806) | Standard Dressing (N=802)
Blisters (Skin and subcutaneous tissue disorders) | 27 (27) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 9 (9) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 14 (14) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was stopped following a planned interim analysis, raising the possibility that it may be underpowered.

The clinical team could not be blinded to the intervention, raising the possibility of bias.

No adjustment was made for multiple comparisons, thus secondary end points could have occurred by chance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03009110/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03009110/ICF_001.pdf